CLINICAL TRIAL: NCT00809484
Title: A Phase III-IV, Multicenter Open Label Trial of Arimidex Alone Versus Arimidex Plus Bisphosphonates in Postmenopausal Patients With Early, Endocrine Positive Breast Cancer.
Brief Title: Arimidex Bone Mass Index and Oral Bisphosphonates
Acronym: ARBI
Status: Completed | Type: Observational
Sponsor: Hellenic Breast Surgeons Society (Other)
Responsible Party: Markopoulos Christos, Hellenic Breast Surgeons Society
Other Study IDs: D5392L0027
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Last update posted 2009-01-06 (Estimated); Status verified 2008-12

CONDITIONS: Breast Cancer; Bone Density
Keywords: Arimidex; Bone Mineral density; Bisphosphonates; Aromatase Inhibitors
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Low risk: Anastrozole 1mg/d, Vit D 400 IU and 500mg Calcium daily
- 2:Moderate risk: Anastrozole 1mg/d, Vit D 400 IU and 500mg Calcium daily, +/- Risedronate 35mg orally once a week
- 3:High risk: Anastrozole 1mg/d, Vit D 400 IU and 500mg Calcium daily, Risedronate 35mg orally once a week

SUMMARY:
To investigate the management of bone health in postmenopausal women with early breast cancer (BCA) scheduled to receive anastrozole. Postmenopausal women with hormone receptor-positive early BCA are assigned to 1 of 3 strata depending on their pre-existing risk of fragility fracture. Patients (pts) with a bone mineral density (BMD) T-score <-2.0 for either spine or hip are designated higher-risk (H) for fracture and receive anastrozole 1 mg/day plus risedronate orally. Moderate-risk (M) pts (T-score <-1.0 for spine or hip but -2.0 at both sites) are randomized to receive anastrozole plus risedronate (A+R) or anastrozole alone. Pts with T-scores -1.0 at both spine and hip were designated lower-risk (L) and receive anastrozole alone. All pts receive calcium and vitamin D. Lumbar spine and total hip BMD are assessed at baseline, 12, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* ER and or PgR positive breast cancer
* Completed Surgery and =/- chemotherapy

Exclusion Criteria:

* metastases
* history of fractures
* HRT or SERMs
* Liver or kidney disfunction

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Posmenopusal women with endocrine responsive breast cancer who are treated with the aromatase inhibitor anastrozole
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2004-05; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hellenic Breast Surgeons Society, Athens, Greece

REFERENCES:
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716
- [Derived] Markopoulos C, Tzoracoleftherakis E, Polychronis A, Venizelos B, Dafni U, Xepapadakis G, Papadiamantis J, Zobolas V, Misitzis J, Kalogerakos K, Sarantopoulou A, Siasos N, Koukouras D, Antonopoulou Z, Lazarou S, Gogas H. Management of anastrozole-induced bone loss in breast cancer patients with oral risedronate: results from the ARBI prospective clinical trial. Breast Cancer Res. 2010;12(2):R24. doi: 10.1186/bcr2565. Epub 2010 Apr 16. PMID 20398352